CLINICAL TRIAL: NCT07268755
Title: Multi-center, Real-world Study on the Treatment of Thoracic Aortic Dissection With a Straight-type Fenestrated Covered Stent System for Thoracic Aortic Aneurysms
Brief Title: Real-world Study on Fenestrated Stent for Thoracic Aortic Dissection
Status: Active, not recruiting | Type: Observational
Sponsor: Qingyou Meng (Other)
Responsible Party: Sponsor-Investigator, Qingyou Meng, Professor, Shanghai General Hospital, China
Organization: Shanghai General Hospital, China (Other)
Other Study IDs: ShanghaiGeneralH
Record Dates: First submitted 2025-11-24; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Thoracic Aortic Dissection; Thoracic Aortic Disease
Keywords: thoracic aortic dissection; Talos; Perforated Stent-Graft
MeSH Terms: conditions — Dissection, Thoracic Aorta

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- TALOS USED GROUP: Population who have received TALOS stents
  Interventions: Device: TALOS

INTERVENTIONS:
Device: TALOS — A Real-World Study on the Effectiveness of the Talos Thoracic Stent Graft System in Thoracic Endovascular Aortic Repair for Aortic Dissection.

SUMMARY:
Study Title:

"Multi-center Real-world Study on Straight Tubular Thoracic Aortic Perforated Stent-Graft System for Treating Thoracic Aortic Dissection"

Purpose:

This study aims to evaluate the effectiveness of the Talos stent-graft system, a new device designed to treat aortic dissection (a life-threatening condition where the inner layer of the aorta tears). The stent has unique features like perforations and tapered design to reduce complications compared to traditional stents.

Key Features of the Talos Stent:

Longer length to cover more of the damaged aorta Perforated design at the distal end to improve blood flow Tapered shape to better match natural aortic anatomy Potentially reduces risks like new tears or spinal cord ischemia

Study Details:

Type: Real-world study (combining prospective and retrospective data) Duration: 3 years (2024-2027) Participants: 320 patients across 5 major hospitals in Shanghai Follow-up: Regular check-ups at 1, 3, 6, 12, and 24 months post-surgery Who Can Participate?

Patients may qualify if they:

Are ≥18 years old Have aortic dissection requiring treatment Have suitable blood vessels for stent placement Can commit to follow-up visits Who Cannot Participate?

Patients with:

Connective tissue disorders (e.g., Marfan syndrome) Active infections or cancer with limited life expectancy Severe allergies to stent materials/contrast dye Pregnancy or planning pregnancy What Does Participation Involve? Pre-Surgery: Physical exams, blood tests, CT scans Surgery: Minimally invasive stent placement via groin artery Post-Surgery: Blood pressure management, antiplatelet medication (e.g., aspirin) Follow-up: CT scans and quality-of-life questionnaires

Potential Benefits:

Improved aortic healing Reduced need for repeat surgeries Better quality of life (measured by VascuQoL questionnaire)

Possible Risks:

Standard stent risks (bleeding, infection, allergic reactions) Device-related complications (leaks, migration, new tears) Organ ischemia (reduced blood flow to kidneys/other organs)

Safety Monitoring:

Independent review of all CT scans 24/7 access to vascular specialists Immediate reporting of any complications

Ethical Protections:

Approved by ethics committees at all hospitals Voluntary participation with signed consent Right to withdraw anytime without affecting care

For Healthcare Providers:

This investigator-initiated study (IIS) is funded by Shanghai Science & Technology Commission. It uses standardized protocols across centers with electronic data capture (EDC) for consistency. The primary endpoint is 12-month treatment success (defined as technical success + no reintervention). Secondary endpoints include aortic remodeling rates and complication profiles.

Contact Information:

Principal Investigator: Dr. Meng Qingyou Institution: Shanghai General Hospital Phone: +86-133-0621-1019

ELIGIBILITY:
Inclusion Criteria:

1. Patients scheduled for or already receiving the Talos stent;
2. Age ≥18 years, any gender, non-pregnant or non-lactating;
3. Diagnosed with aortic dissection;
4. Presence of a ≥15mm effective proximal landing zone;
5. Having eligible access artery anatomy;
6. Expected survival >1 year;
7. Capable of understanding the trial purpose, voluntarily participating, signing informed consent, and willing to undergo follow-up.

Exclusion Criteria

1. Definitive diagnosis of aortic-related connective tissue disorders (e.g., Marfan syndrome);
2. Subjects with infectious aortic dissection;
3. Documented allergy to nitinol alloys, contrast agents, or related materials;
4. Severe hepatic/renal dysfunction (ALT or AST >2.5×ULN, serum creatinine >2×ULN);
5. Uncontrolled severe infections (e.g., bacteremia or septicemia);
6. History of active bleeding, coagulopathy, or refusal of blood transfusion;
7. Malignancy with life expectancy <1 year;
8. Pregnancy, lactation, or planned pregnancy during the trial;
9. Concurrent participation in other drug/device trials without completing primary endpoints;
10. Poor compliance with anticipated inability to complete follow-up;
11. Other investigator-determined contraindications for endovascular therapy (e.g., unsuitable vascular access, non-cooperation).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: a group with Thoracic Aortic Dissection
Sampling Method: Non-Probability Sample
Enrollment: 320 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Treatment success rate at 12 months post-procedure | 12 months
  Defined as immediate technical success after the procedure and no reintervention required during the 12-month follow-up period.
Treatment success rate at 12 months post-procedure, defined as immediate technical success after the procedure and no reintervention required during the 12-month follow-up period. | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Jiaotong University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes